CLINICAL TRIAL: NCT00024206
Title: A Phase I Surrogate Endpoint Trial of SU6668 in Patients With Incurable Solid Tumors
Brief Title: SU6668 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02412; ID00-184; U01CA062461 (NIH); CDR0000068900 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-09-13; First posted 2003-10-21 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — orantinib

ARMS (1):
- Treatment (orantinib) (Experimental): Patients receive oral SU6668 twice daily on days 1-28. Courses repeat every 4 weeks in the absence of unacceptable toxicity or disease progression of 100% or more.
  Cohorts of at least 6 patients receive escalating doses of SU6668 until the OBD is determined. Once the OBD is reached, dose escalation continues until the maximum tolerated dose (MTD) is determined (if possible). The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: orantinib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: orantinib — Given orally
  Other Names: SU006668; SU6668; Sugen SU6668; TSU 68
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effectiveness of SU6668 in treating patients who have advanced solid tumors. SU6668 may stop the growth of solid tumors by stopping blood flow to the tumor

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the optimal biologically effective dose of SU6668 in patients with advanced solid tumors.

II. Assess the safety and tolerability of this therapy in these patients. III. Determine the pharmacokinetic profile and interpatient pharmacologic variability of this therapy in these patients.

IV. Determine the extent, frequency, and duration of any tumor responses in patients treated with this therapy.

V. Determine a recommended phase II dose of SU6668 for future clinical studies.

OUTLINE: This is a dose-escalation study.

Patients receive oral SU6668 twice daily on days 1-28. Courses repeat every 4 weeks in the absence of unacceptable toxicity or disease progression of 100% or more.

Cohorts of at least 6 patients receive escalating doses of SU6668 until the optimal biologically effective dose (OBD) is determined. Once the OBD is reached, dose escalation continues until the maximum tolerated dose (MTD) is determined (if possible). The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumor for which no standard therapy exists
* At least 1 measurable tumor lesion (at least 2 cm) not previously irradiated
* No history of brain metastases

  * Negative brain CT/MRI required for patients with signs and symptoms suspicious for brain metastases
* Performance status - ECOG 0-1
* WBC greater than 3,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL
* No history of bleeding diathesis
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT less than 2.5 times ULN
* Creatinine less than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min
* No concurrent uncontrolled medical or psychiatric disorders
* No severe iodine allergy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 30 days since prior over-the-counter, anticancer biologic agents (e.g., shark cartilage)
* No concurrent over-the-counter, anticancer biologic agents (e.g., shark cartilage)
* At least 3 weeks since prior cytotoxic or cytostatic agents (6 weeks for nitrosoureas or mitomycin)
* Patients with ECOG performance status 0:

  * Any number of prior chemotherapy regimens allowed
* Patients with ECOG performance status 1:

  * No more than 3 prior chemotherapy regimens for metastatic or recurrent disease
  * The same drug given on a different schedule does not count as a different regimen
  * Prior adjuvant chemotherapy for non-metastatic disease or as part of a concurrent chemoradiotherapy protocol is allowed but does not count as part of the 3-regimen limit
* See Disease Characteristics
* See Chemotherapy
* At least 3 weeks since prior radiotherapy to nonindicator lesions
* No concurrent radiotherapy
* At least 24 hours since prior minor surgery (e.g., central venous catheter placement)
* At least 4 weeks since prior major surgery (e.g., laparotomy, thoracotomy, or craniotomy)
* At least 30 days since prior anticancer herbal remedies
* At least 30 days since prior investigational agents
* No concurrent anticancer herbal remedies
* No other concurrent investigational or anticancer medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2001-07; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, as defined by the Coding Symbols for a Thesaurus of Adverse Reaction Terms (COSTART) term and body system, graded according to the National Cancer Institute Common Toxicity Criteria v2.0 | Up to 2 years
Maximally tolerated dose of orantinib, graded according to the NCI CTC v2.0 | Up to 4 weeks

SECONDARY OUTCOMES:
Tumor response, assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 2 years
Angiogenic surrogate measures in terms of change in cytokines over time | Days 8, 15, and 22
  A mixed-effects analysis of variance (ANOVA) model will be used, and a fixed-effects model in which the same polynomial is fit for each patient will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Herbst, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States